CLINICAL TRIAL: NCT00525759
Title: A Randomised Phase II Feasibility Study Investigating the Biological Effects of the Addition of Zoledronic Acid to Neoadjuvant Combination Chemotherapy on Invasive Breast Cancer
Brief Title: Investigating the Biological Effects of the Addition of Zoledronic Acid to Pre-operative Chemotherapy in Breast Cancer
Acronym: ANZAC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Director of Research & Development, Sheffield Teaching Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH14707
Record Dates: First submitted 2007-09-05; First posted 2007-09-06 (Estimated); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Zoledronic acid; Neoadjuvant chemotherapy; Synergy; Apoptosis
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluorouracil; Epirubicin; Cyclophosphamide; Docetaxel; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Neoadjuvant chemotherapy alone
  Interventions: Drug: 5-FU, Epirubicin, Cyclophosphamide, Docetaxel
- B (Experimental): Neoadjuvant chemotherapy + zoledronic acid
  Interventions: Drug: 5-FU, Epirubicin, Cyclophosphamide, Docetaxel, Zoledronic acid

INTERVENTIONS:
Drug: 5-FU, Epirubicin, Cyclophosphamide, Docetaxel — 3 cycles of FEC q3w, followed by 3 cycles of docetaxel q3w FEC: 5FU 500mg/m2 intravenous bolus D1, Epirubicin 100mg/m2 intravenous bolus D1, Cyclophosphamide 500mg/m2 intravenous bolus D1) every 21 days Docetaxel: (100mg/ m2 intravenous infusion) every 21 days
  Arms: A
Drug: 5-FU, Epirubicin, Cyclophosphamide, Docetaxel, Zoledronic acid — 3 cycles of FEC q3w, followed by 3 cycles of docetaxel q3w FEC: 5FU 500mg/m2 intravenous bolus D1, Epirubicin 100mg/m2 intravenous bolus D1, Cyclophosphamide 500mg/m2 intravenous bolus D1) every 21 days Docetaxel: (100mg/ m2 intravenous infusion) every 21 days Zoledronic acid: 4mg intravenous infusion Day 2, AFTER FIRST CYCLE CHEMOTHERAPY ONLY
  Arms: B

SUMMARY:
There is clear preclinical in vitro and in vivo evidence of sequence dependent synergy between chemotherapy agents and zoledronic acid. The aim of the study is to investigate if the synergistic increase in tumour cell apoptosis observed in preclinical studies occurs in patients. The hypothesis for this study is that there may be anti-tumour benefits of the sequential application of chemotherapy agents followed by zoledronic acid in patients with invasive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with histological diagnosis of invasive breast cancer requiring neoadjuvant chemotherapy
* T2 tumour or above
* WHO Performance status of 0,1 or 2
* Must consent to or have undergone a core biopsy for diagnosis of breast cancer AND consent to undergo an additional core biopsy prior to the second cycle of chemotherapy (Day 5 +/- Day 21)
* Written informed consent

Exclusion Criteria:

* Previous chemotherapy or radiotherapy to treated breast
* Evidence of metastatic disease or recurrent breast cancer or previous malignancy (some exceptions)
* Calculated creatinine clearance < 40mls/min
* Prior treatment with bisphosphonates in last year or known contraindications to bisphosphonate therapy
* Concurrent tamoxifen or aromatase inhibitor medication
* Pregnant or lactating women
* Cardiac dysfunction that precludes use of anthracycline chemotherapy
* Unwilling to have extra interim biopsy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-07; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Increase in apoptotic index between diagnostic core biopsy and repeat core biopsy taken on day 5 | Repeat biopsy on day 5 (+/- day 21)

SECONDARY OUTCOMES:
Reduction in Ki67 immunostaining between preoperative core biopsy, repeat core biopsy on day 5, +/- day 21, and operative specimen | Day 5, +/- Day 21, surgical specimen
Changes in serum angiogenesis markers between pre-treatment and operative time points | Pre-treatment, Day 5, day 21, pre-surgery
Changes in bone biochemical markers between pre-treatment, treatment and operative timepoints | Pre-treatment, Day 5, day 21, pre-surgery
Detection of, and changes in, circulating tumour cells in peripheral blood taken pre-treatment, during treatment and following treatment | Pre-treatment, day 5, day 21, pre-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Coleman, MB BS, MD, Principal Investigator — Academic Unit of Clinical Oncology, University of Sheffield
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust / Weston Park Hospital, Sheffield, South Yorkshire, United Kingdom

REFERENCES:
- [Background] Jagdev SP, Coleman RE, Shipman CM, Rostami-H A, Croucher PI. The bisphosphonate, zoledronic acid, induces apoptosis of breast cancer cells: evidence for synergy with paclitaxel. Br J Cancer. 2001 Apr 20;84(8):1126-34. doi: 10.1054/bjoc.2001.1727. PMID 11308265
- [Background] Neville-Webbe HL, Rostami-Hodjegan A, Evans CA, Coleman RE, Holen I. Sequence- and schedule-dependent enhancement of zoledronic acid induced apoptosis by doxorubicin in breast and prostate cancer cells. Int J Cancer. 2005 Jan 20;113(3):364-71. doi: 10.1002/ijc.20602. PMID 15455384
- [Background] Ottewell PD, Jones M, Coleman RE, Holen I. Synergistic effects of cytotoxic drugs and anti-resorptive agents in vitro and in vivo. In 29th Annual San Antonio Breast Cancer Symposium Vol.100 Suppl.1 Abstract 6102, Breast Cancer Research and Treatment
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Winter MC, Wilson C, Syddall SP, Cross SS, Evans A, Ingram CE, Jolley IJ, Hatton MQ, Freeman JV, Mori S, Holen I, Coleman RE. Neoadjuvant chemotherapy with or without zoledronic acid in early breast cancer--a randomized biomarker pilot study. Clin Cancer Res. 2013 May 15;19(10):2755-65. doi: 10.1158/1078-0432.CCR-12-3235. Epub 2013 Mar 20. PMID 23515409